CLINICAL TRIAL: NCT06469073
Title: Ultrasound-guided Modified Transversus Thoracic Muscle Plane Block and Erector Spinal Muscle Plane Block in Heart Valve Replacement Surgery With Median Incision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Le Yu (Other)
Responsible Party: Sponsor-Investigator, Le Yu, Clinicians, Shanghai East Hospital of Tongji University
Organization: Shanghai East Hospital of Tongji University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024.6.25-2024.8.25
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transversus thoracic muscle plane block (T) group (Experimental)
  Interventions: Procedure: Transversus thoracic muscle plane block or Erector spinal plane block
- Erector spinal plane block (E) group (Experimental)
  Interventions: Procedure: Transversus thoracic muscle plane block or Erector spinal plane block
- General anesthesia only (G) group (No Intervention)

INTERVENTIONS:
Procedure: Transversus thoracic muscle plane block or Erector spinal plane block — Transversus thoracic muscle plane block or Erector spinal plane block
  Arms: Erector spinal plane block (E) group; Transversus thoracic muscle plane block (T) group

SUMMARY:
Sternum midline incision can offer better view under open-heart surgery and bigger operating space, and therefore it has been widely used in most cardiac surgery. If an event of urgency occurs, it takes on a more important role than infrasternal small incision. However, sternum midline incision may cause serious pain and aggravates stress response, and therefore patients are often reluctant to cooperate to cough which exerts adverse effect on postoperative rehabilitation, and even causes serious complications such as pulmonary inflammation, myocardial infarction and heart failure. Thus, the relief of pain and better perioperative analgesia are very important for these patients. Transversus thoracic muscle plane(TTMP) block and erector spinal muscle plane(ESP) block are used in open heart surgery currently, and they can provide good analgesia. This study aimed to investigate the hemodynamic stability, total amount of analgesic use, perioperative pain, stress response, postoperative complication and recovery in patients receiving TMP and ESP.

ELIGIBILITY:
Inclusion Criteria:

* patients (18-75 years) with BMI at 18-25 kg/m2, ASA Ⅱ- Ⅲ and NYHA Ⅱ-Ⅲ who scheduled to undergo mitral valve or aortic valve replacement surgery.

Exclusion Criteria:

* a second operation, preoperative ejection fraction (EF) < 40%, complicated coronary heart disease, intra-aortic balloon counterpulsation (IABP) support, psychiatric abnormalities, history of allergy to anesthetic drugs, liver or kidney dysfunction, coagulation abnormality, endocrine system diseases and metabolic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-25 (Estimated); Primary Completion 2024-08-25 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure | entering the operating room (T0)
  an average blood pressure in an individual during a single cardiac cycle
Mean arterial pressure | intubation (T1)
  an average blood pressure in an individual during a single cardiac cycle
Mean arterial pressure | skin incision (T2)
  an average blood pressure in an individual during a single cardiac cycle
Mean arterial pressure | breast opening (T3)
  an average blood pressure in an individual during a single cardiac cycle
Mean arterial pressure | sternal retractor placement (T4)
  an average blood pressure in an individual during a single cardiac cycle
Mean arterial pressure | pericardium incision (T5)
  an average blood pressure in an individual during a single cardiac cycle
Mean arterial pressure | steel wire pulling (T6)
  an average blood pressure in an individual during a single cardiac cycle
Heart beats | entering the operating room (T0)
  the number of times each minute that heart beats
Heart beats | intubation (T1)
  the number of times each minute that heart beats
Heart beats | skin incision (T2)
  the number of times each minute that heart beats
Heart beats | breast opening (T3)
  the number of times each minute that heart beats
Heart beats | sternal retractor placement (T4)
  the number of times each minute that heart beats
Heart beats | pericardium incision (T5)
  the number of times each minute that heart beats
Heart beats | steel wire pulling (T6)
  the number of times each minute that heart beats

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital of Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided